CLINICAL TRIAL: NCT01832324
Title: Molecular Basis of Food Allergy and Food Tolerance
Brief Title: Molecular Basis of Food Allergy
Status: Enrolling by invitation | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 08-005998
Record Dates: First submitted 2013-04-12; First posted 2013-04-16 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Food Allergy; Eosinophilic Esophagitis
Keywords: Food Allergy; Eosinophilic Esophagitis; Food Protein Induced Enterocolitis; iNKT Cells; T cells
MeSH Terms: conditions — Food Hypersensitivity; Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, sera and PBMC
Oversight: Data Monitoring Committee: No

SUMMARY:
The Study examines the molecular basis of food allergy. It explores the interaction between T cells, InKT cells, basophils and cytokines in the development of food allergy. The study also explores these factors in development of tolerance "outgrowing" food allergy. It will also explore the genetic factors that lead to the development of food allergy.

The study examines all type of food allergy including IgE mediated reactions, Eosinophilic Esophagitis and Food Protein Induced Enterocolitis

DETAILED DESCRIPTION:
Food Allergy (FA) is a common pediatric atopic disease. Characteristically children affected by FA become sensitized to food in the first few months of life and spontaneously outgrow the disease by 5-6 years of age in about 80% of cases. At the present time, diagnosis of FA is made by a combination of history, skin testing and food challenge. The pathogenic mechanisms leading to food sensitization and subsequent spontaneous tolerance development are not understood.

ELIGIBILITY:
Inclusion Criteria for Study Group:

1. Males or females age 1 month to 65 years.
2. Diagnosis of Food Allergy. Food Allergy can be either IgE or non-IgE mediated food allergy including Eosinophilic Esophagitis and Food Protein Induced Enterocolitis.

Inclusion Criteria for Control group:

1. Age and sex matched patients without food allergies
2. Sibling and parents of patients with food allergies

Inclusion Criteria for Control group with atopy:

1. Age and sex matched patients without food allergies
2. Sibling and parents of patients with food allergies
3. Patients with atopy

Exclusion Criteria

1. Underlying disease or medical problem that is judged to serious or risky to allow 3 ml/kg of blood to be drawn from a vein (such as serious anemia, cancer, poor vein abscess, serious infections).
2. Subjects that do not meet the enrollment criteria may not be enrolled. Any violations of these criteria will be reported in accordance with Institutional Review Board (IRB) policies and procedures study procedures.

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Food Allergy (Both IgE and Non-IgE Mediated) Atopic Controls Healthy controls
Sampling Method: Probability Sample
Enrollment: 5300 (Estimated)
Dates: Start 2011-01; Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Blood sample for mechanistic studies: | 1 year
  Blood will be obtained by venipuncture. The blood samples will be used to estimate the frequency of to estimate the frequency and the products of cells involved in the allergic reaction. We will quantify the number of lymphocytes and their subsets, and the number granulocytes (neutrophils, basophils, and eosinophils) and monocytes and we will analyze their products (such as cytokines, chemokines, prostanoids). Such analysis will be performed doing cytoflow studies, using 4 color flow cytometry (BD FACSCalibur Flow XCytometry System) at the Children's Hospital Flow Cytometry core facilities, ELISA, mRNA analysis and western blots using when indicated the Nucleic Acid/Protein Core. If blood won't be all used up in the aforementioned tests it will be stored in nitrogen liquid for future similar tests or repetition of the ones already performed in case of technical problem with the first attempt.
Blood sample for genetic study (optional) | 1 year
  The Center for Applied Genomics (CAG) will perform genetic analysis. All subjects (cases and controls) have been or will be genotyped on the Illumina HumanHap BeadArray SNP platform, and data has been stored in following an IRB approved protocol
  Whole Exon Sequencing (also known as targeted exome capture) is an efficient strategy to selectively sequence the coding regions of the genome as a cheaper but still effective alternative to whole genome sequencing. Exons are short, functionally important sequences of DNA which represent the regions in genes that are translated into protein and the untranslated region flanking them (UTR). It is estimated that the protein coding regions of the human genome constitute about 85% of the disease-causing mutations.
  Statistical analysis will be done in conjunction with CAG and Children's Hospital of Philadelphia (CHOP) bioinformatics center. We will compare the genetic variants identified between sequencing and SNPs -based genotyping.
EndoPat Test (optional) | 1 year
  EndoPat is a noninvasive endothelial function assessment. Patient should rest comfortably for 10 minutes prior to the test. Using a standard blood pressure cuff, the brachial artery is occluded for a 5 minute period. When the cuff is released, EndoPat measures blood flow rates pre-occlusion and post-occlusion. This test requires patients to sit still for 15 minutes. It's recommended that the patient fast 3 to 8 hours before the test. In addition, the following drugs should not be used for 24 hours before testing: Nitroglycerine, Alpha-blockers, beta-blockers, and calcium channel blockers, ACE inhibitors, Statins

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Spergel, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Deidentiifed data including specific IgE, results of basophil assay and what individual food that the patient is reacting to will be included.

REFERENCES:
- [Background] Ruffner MA, Zhang Z, Maurer K, Muir AB, Cianferoni A, Sullivan KE, Spergel JM. RNA sequencing identifies global transcriptional changes in peripheral CD4+ cells during active oesophagitis and following epicutaneous immunotherapy in eosinophilic oesophagitis. Clin Transl Immunology. 2021 Jul 22;10(7):e1314. doi: 10.1002/cti2.1314. eCollection 2021. PMID 34322233
- [Background] Dilollo J, Rodriguez-Lopez EM, Wilkey L, Martin EK, Spergel JM, Hill DA. Peripheral markers of allergen-specific immune activation predict clinical allergy in eosinophilic esophagitis. Allergy. 2021 Nov;76(11):3470-3478. doi: 10.1111/all.14854. Epub 2021 May 14. PMID 33840099